CLINICAL TRIAL: NCT00794040
Title: A Controlled Trial of Citalopram Added to Methylphenidate in Youth With Severe Mood Dysregulation
Brief Title: A Controlled Trial of Serotonin Reuptake Inhibitors Added to Stimulant Medication in Youth With Severe Mood Dysregulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 090034; 09-M-0034
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2018-02-01

CONDITIONS: Mood Disorder; Mental Disorder Diagnosed in Childhood; Attention Deficit and Disruptive Behavior Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Irritability; Attention Deficit Hyperactivity Disorder; Explosive; Tantrums; Bipolar Mood Disorder; Mood Disorder; Childhood Mood Disorder; ADHD
MeSH Terms: conditions — Mood Disorders; Attention Deficit Disorder with Hyperactivity; Attention Deficit and Disruptive Behavior Disorders; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Add-on citalopram following optimized methylphenidate (Active Comparator): After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram or placebo
  Interventions: Drug: Add-on citalopram following optimized methylphenidate
- Add-on placebo after optimized methylphenidate (Placebo Comparator): After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram or placebo
  Interventions: Drug: Add-on placebo following optimized methylphenidate

INTERVENTIONS:
Drug: Add-on citalopram following optimized methylphenidate — After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram or placebo
  Arms: Add-on citalopram following optimized methylphenidate
Drug: Add-on placebo following optimized methylphenidate — After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram or placebo
  Arms: Add-on placebo after optimized methylphenidate

SUMMARY:
Severe mood dysregulation (SMD) is a very common syndrome in children. Its symptoms include very severe irritability, including persistent anger and frequent outbursts, as well as distractibility, hyperactivity, and other symptoms of attention deficit hyperactivity disorder (ADHD). Many children with SMD receive the diagnosis of bipolar disorder (BD) in the community, although they do not have clear manic episodes (with symptoms such as extreme happiness and decreased need for sleep). Because SMD has not been studied in depth, we do not know which medications are most helpful to those with SMD. This study will evaluate the effectiveness of the stimulant medication methylphenidate (MPH, more commonly known as Ritalin ) when combined (or not combined) with the antidepressant citalopram (Celexa ) in treating symptoms of SMD in children and adolescents. This study will provide information about how to treat SMD in youth.

This study will include approximately 80 patients between 7 and 17 years of age with SMD. The patient s symptoms must have started before age 12.

The study will consist of four phases carried out over 4 to 5 months. During Phase 1, the patient will undergo blood and urine tests, and will gradually taper off his or her medication. The duration of this phase depends on the patient s medication before starting the study. In Phase 2, the patient remains off all medication for 1 week. In Phase 3, the patient will be treated with MPH for 2 weeks, and then will be randomly assigned to receive either MPH plus citalopram or MPH plus a placebo for a further 8 weeks. In Phase 4, the researchers will evaluate the effectiveness of the medications taken, and begin an open treatment phase using medications that they deem appropriate for that patient (this may include MPH with citalopram and/or other medication combinations).

Most patients will be admitted to the Pediatric Behavioral Health Unit at the National Institutes of Health Clinical Center during the medication withdrawal part of the study (Phases 1 and 2). From Phase 3 on, a patient may participate as an inpatient, outpatient, or in day treatment, depending on what is in his or her best interests.

...

DETAILED DESCRIPTION:
Objective: To test the efficacy of citalopram plus methylphenidate vs. placebo plus methylphenidate in decreasing irritability in youth with severe mood dysregulation.

Study population: Youth ages 7-17 with severe mood dysregulation (SMD). SMD is characterized by nonepisodic, impairing irritability (defined as increased reactivity to negative emotional stimuli at least 3 times/week and angry or sad mood, most days, most of the time, noticeable to others) and hyperarousal (three of: distractibility, intrusiveness, pressured speech, racing thoughts, agitation, insomnia), with onset before age 12. Many of these children receive the diagnosis of bipolar disorder (BD) in the community, although they do not meet DSM-IV criteria for BD because of the lack of distinct manic episodes.

Design: Medication withdrawal, followed by a 5-week dose stabilization phase of methylphenidate and an 8-week double-blind, placebo-controlled treatment trial of citalopram plus methylphenidate vs. placebo plus methylphenidate. There will also be optional open treatment at the end, so that all patients have the opportunity to have a total of up to 10 weeks of citalopram plus methylphenidate. The target dose of citalopram will be 20-40 mg/day.

Outcome measures: The primary outcome measures will be the Aberrant Behavior Checklist Irritability subscale and the CGI-I.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Ages 7-17
  2. Abnormal mood (specifically, anger, sadness, and/or irritability), present at least half of the day most days, and of sufficient severity to be noticeable by people in the child s environment (e.g. parents, teachers, peers).
  3. Hyperarousal, as defined by at least three of the following symptoms: insomnia, agitation, distractibility, racing thoughts or flight of ideas, pressured speech, intrusiveness
  4. Compared to his/her peers, the child exhibits markedly increased reactivity to negative emotional stimuli that is manifest verbally and/or behaviorally. For example, the child responds to frustration with extended temper tantrums (inappropriate for age and/or precipitating event), verbal rages, and/or aggression toward people or property. Such events occur, on average, at least three times a week
  5. Criteria 2, 3, and 4 are currently present and have been present for at least 12 months without any symptom-free periods exceeding two months.
  6. The onset of symptoms must be prior to age 12 years.
  7. The symptoms are severe in at least one setting (e.g. violent outbursts, extreme verbal abuse, assaultiveness at home, school, or with peers). In addition, there are at least mild symptoms (distractibility, intrusiveness) in a second setting.
  8. Currently in treatment with a psychiatrist for the symptoms.
  9. The child is failing his/her treatment. To meet this criterion:

     i.The child s current CGAS score must be less than or equal to 60.

     ii.The child s psychiatrist/treater must agree that the child s response to his/her current treatment is no more than minimal. According to this criterion, it would be clinically appropriate to change the child s current treatment.

     iii.On the basis of record review and interviews with child and parent, the research team agrees that the child s response to his/her current treatment is no more than minimal.

     iv.The child has a score of greater than 12 on the irritability subscale of the Aberrant Behavior Checklist.

     EXCLUSION CRITERIA:

  <!-- -->

  1. As assessed in the mania section of the K-SADS-PL, the individual exhibits any of these cardinal bipolar symptoms in distinct periods lasting more than 1 day, and therefore meets criteria for bipolar disorder not otherwise specified:

     i) Elevated or expansive mood

     ii) Grandiosity or inflated self-esteem

     iii) Decreased need for sleep

     iv) Increase in goal-directed activity (this can result in the excessive involvement in pleasurable activities that have a high potential for painful consequences)
  2. Meets criteria for schizophrenia, schizophreniform disorder, schizoaffective illness, more than mild PDD, or PTSD.
  3. Meets criteria for substance use disorder in the three months prior to randomization.
  4. IQ less than 70
  5. The symptoms are due to the direct physiological effects of a drug of abuse, or to a general medical or neurological condition.
  6. Currently pregnant or lactating, or sexually active without using a barrier method of contraception.
  7. Failed an adequate trial (defined as four weeks of consecutive treatment at the minimally effective) or severe ill effects while on citalopram (at least 20 mg) or escitalopram (at least 10 mg).
  8. Hypersensitivity or severe adverse reaction to methylphenidate
  9. A history of serious adverse reactions (psychosis, severely increased activation compared to baseline) to methylphenidate or amphetamines.
  10. Any chronic medical condition that requires medications that are contraindicated with SSRIs or methylphenidate, or any serious chronic or unstable medical disorder.
  11. Medical contraindications to treatment with SSRI or stimulant (e.g. liver, seizure, renal, platelet disorder).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2008-11-17; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argyris Stringaris, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amsterdam JD, Shults J. Comparison of fluoxetine, olanzapine, and combined fluoxetine plus olanzapine initial therapy of bipolar type I and type II major depression--lack of manic induction. J Affect Disord. 2005 Jul;87(1):121-30. doi: 10.1016/j.jad.2005.02.018. PMID 15923042
- [Background] Baumer FM, Howe M, Gallelli K, Simeonova DI, Hallmayer J, Chang KD. A pilot study of antidepressant-induced mania in pediatric bipolar disorder: Characteristics, risk factors, and the serotonin transporter gene. Biol Psychiatry. 2006 Nov 1;60(9):1005-12. doi: 10.1016/j.biopsych.2006.06.010. Epub 2006 Aug 30. PMID 16945343
- [Background] Binks CA, Fenton M, McCarthy L, Lee T, Adams CE, Duggan C. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005653. doi: 10.1002/14651858.CD005653. PMID 16437535
- [Derived] Towbin K, Vidal-Ribas P, Brotman MA, Pickles A, Miller KV, Kaiser A, Vitale AD, Engel C, Overman GP, Davis M, Lee B, McNeil C, Wheeler W, Yokum CH, Haring CT, Roule A, Wambach CG, Sharif-Askary B, Pine DS, Leibenluft E, Stringaris A. A Double-Blind Randomized Placebo-Controlled Trial of Citalopram Adjunctive to Stimulant Medication in Youth With Chronic Severe Irritability. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):350-361. doi: 10.1016/j.jaac.2019.05.015. Epub 2019 May 23. PMID 31128268
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-M-0034.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at the National Institute of Mental Health Division of Intramural Research Programs (NIMH DIRP) from November 2008 until January 2018. The inpatient part of the study took place at the Child Psychiatric Unit of the NIH Clinical Center.
Pre-assignment Details: Enrolled participants (N=103) went through a medication wash-out period. n=22 participants withdrew assent before or during this period, and 12 participants met exclusion criteria. Then 69 participants began methylphenidate optimization; of those, 4 withdrew assent, 12 did not meet inclusion criteria. n=53 were randomized, and 49 analyzed.
Groups:
- Add-on Citalopram Following Optimized Methylphenidate: After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram (this arm) or placebo
- Add-on Placebo Following Optimized Methylphenidate: After optimized treatment with methylphenidate, those who meet threshold for chronic irritability are randomized to add-on citalopram or placebo (this arm)
Period: Overall Study
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Started | 25 | 28
Completed | 22 | 23
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Whereas 53 participants were randomized, 49 participants were analyzed using intent-to-treat analysis. The first 4 participants recruited were excluded because a different version of the primary outcome measure (i.e., CGI) was collected in these participants and therefore was not comparable to the remaining participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.5) | 11.7 (2.1) | 11.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 13 | 20 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 19 | 20 | 39
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 26 | 49
Clinical Global Impression - Severity (CGI-S) collected at Admission [Mean (Standard Deviation); unit: units on a scale] — A measure of severity of irritability scale (from 1=Normal, not at all ill to 7=Among the most extremely ill patients). Two graduate-level, highly-experienced clinicians completed weekly the CGI, with child and parent/nursing staff as a source of information. Ratings were reached by consensus in a case conference with a senior child and adolescent psychiatrist (KT); all clinicians and participants were blind to the treatment condition.
  units on a scale | 4.4 (0.6) | 4.6 (0.5) | 4.5 (0.5)
Children's Global Assessment of Severity (CGAS) collected at Admission [Mean (Standard Deviation); unit: units on a scale] — A measure of overall functional impairment with scores ranging from 1=Most impaired to 100=Not impaired at all.
  units on a scale | 44 (6.1) | 41.7 (2.2) | 42.8 (4.5)
Children's Depression Rating Scale (CDRS) collected at Admission [Mean (Standard Deviation); unit: units on a scale] — A measure of depressive symptoms severity ranging 17-113, where scores >40 are considered over the clinical threshold, and scores <28 are considered within the healthy range.
  units on a scale | 29.7 (5.9) | 32.0 (7.6) | 30.1 (6.9)
Pediatric Anxiety Rating Scale (PARS) collected at Admission [Mean (Standard Deviation); unit: units on a scale] — A measure of anxiety symptoms severity with scores ranging 0-25. Higher values represent a worse outcome.
  units on a scale | 15.7 (4.5) | 14.8 (4.7) | 15.1 (4.8)
Psychiatric disorders information collected at Admission using the K-SADS-PL [Count of Participants; unit: Participants] — Presence of co-occurring psychiatric disorders at the time of enrollment to study measured with a semi-structured interview, the Kiddie Schedule for Affective Disorders Present and Lifetime Version (K-SADS-PL).
  Participants
    Any disorder | 23 | 26 | 49
    Attention Deficit Hyperactivity Disorder | 20 | 24 | 44
    Oppositional Defiant Disorder | 17 | 22 | 39
    Conduct Disorder | 0 | 1 | 1
    Any Anxiety disorder | 13 | 15 | 28
Clinical Global Impression - Severity (CGI-S) collected before Randomization [Mean (Standard Deviation); unit: units on a scale] — A measure of severity of irritability scale (from 1=Normal, not at all ill to 7=Among the most extremely ill patients). Two graduate-level, highly-experienced clinicians completed weekly the CGI, with child and parent/nursing staff as a source of information. Ratings were reached by consensus in a case conference with a senior child and adolescent psychiatrist (KT); all clinicians and participants were blind to the treatment condition.
  units on a scale | 4.0 (0.5) | 4.3 (0.6) | 4.2 (0.6)
Children's Global Assessment of Severity (CGAS) collected before Randomization [Mean (Standard Deviation); unit: units on a scale] — A measure of overall functional impairment with scores ranging from 1=Most impaired to 100=Not impaired at all
  units on a scale | 44.4 (3.3) | 42.9 (3.6) | 43.6 (3.5)
Children's Depression Rating Scale (CDRS) collected before Randomization [Mean (Standard Deviation); unit: units on a scale] — A measure of depressive symptoms severity ranging 17-113, where scores >40 are considered over the clinical threshold, and scores <28 are considered within the healthy range
  units on a scale | 29.4 (5.7) | 34.6 (8.6) | 32.1 (7.7)
Pediatric Anxiety Rating Scale (PARS) collected before Randomization [Mean (Standard Deviation); unit: units on a scale] — A measure of anxiety symptoms severity with scores ranging 0-25. Higher values represent a worse outcome.
  units on a scale | 13.3 (5.9) | 15.8 (5.2) | 14.8 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That "Much Improved" (Score of 2) in, or "Completely Recovered" (Score of 1) From Their Irritability Severity, as Measured With the Clinical Global Impression-Improvement (CGI-I).
Description: A measure of change of irritability severity taking the baseline before randomization as a reference. Scores range 1 to 8, in which 1=Completely recovered,... 5=Unchanged,... 8=Much worse.
  Percentage of participants who responded are based on an estimation and might not match exactly with discrete numbers of participants based on the denominator.
Time Frame: Collected weekly during the 8-week trial. The 8th-week outcome is reported.
Population: as for baseline characteristics
Measure: Number; unit: estimated percentage of participants
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Number analyzed (Participants) | 23 | 26
estimated percentage of participants | 35 | 6
Statistical Analysis 1: Comparison: Add-on Citalopram Following Optimized Methylphenidate vs Add-on Placebo Following Optimized Methylphenidate; Test type: Superiority; p = 0.006, Multilevel growth curve model — priori threshold p<0.05; Odds Ratio (OR) = 11.7, 95% CI 2-sided [2.00 to 68.16]

2. Secondary Outcome: Irritability Severity at 8th Week of Trial.
Description: Clinical Global Impression-Severity (CGI-S): A measure of severity of irritability scale (from 1=Normal, not at all ill to 7=Among the most extremely ill patients).
Time Frame: Collected weekly during the 8th week trial. The 8th-week outcome is reported.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Number analyzed (Participants) | 23 | 26
units on a scale | 3.1 (0.3) | 3.9 (0.3)
Statistical Analysis 1: Comparison: Add-on Citalopram Following Optimized Methylphenidate vs Add-on Placebo Following Optimized Methylphenidate; Test type: Superiority; p = 0.085, Multilevel growth curve model — priori threshold <0.05; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.32 to 0.09]

3. Secondary Outcome: Functional Impairment at 8th Week of Trial
Description: Difference in functional impairment at 8th week of trial as measured with Children's Global Impression Scale (CGAS) with scores ranging from 1=Most impaired to 100=Not impaired at all.
Time Frame: Collected weekly during the 8th week trial. The 8th-week outcome is reported.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Number analyzed (Participants) | 23 | 26
units on a scale | 52.6 (2.3) | 47.2 (2.1)
Statistical Analysis 1: Comparison: Add-on Citalopram Following Optimized Methylphenidate vs Add-on Placebo Following Optimized Methylphenidate; Test type: Superiority; p = 0.124, Wilcoxon (Mann-Whitney) — priori threshold p<0.05; Mean Difference (Final Values) = 4.72, 95% CI 2-sided [-1.30 to 10.74]

4. Secondary Outcome: Depressive Symptoms at 8th Week of Trial
Description: Difference in depressive symptoms at 8th week of trial as measured with Children's Depression Rating Scale (CDRS) with scores ranging 17-113, where scores >40 are considered over the clinical threshold, and scores <28 are considered within the healthy range.
Time Frame: Collected weekly during the 8th week trial. The 8th-week outcome is reported.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Number analyzed (Participants) | 23 | 26
units on a scale | 28.6 (1.8) | 30.1 (1.8)
Statistical Analysis 1: Comparison: Add-on Citalopram Following Optimized Methylphenidate vs Add-on Placebo Following Optimized Methylphenidate; Test type: Superiority; p = 0.993, Multilevel growth curve model — priori threshold p<0.05; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-4.76 to 4.80]

5. Secondary Outcome: Anxiety Symptoms at 8th Week of Trial
Description: Difference in anxiety symptoms at 8th week of trial as measured with the Pediatric Anxiety Rating Scale (PARS) with scores ranging 0-25. Higher values represent a worse outcome.
Time Frame: Collected weekly during the 8th week trial. The 8th-week outcome is reported.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
Number analyzed (Participants) | 23 | 26
units on a scale | 12.0 (1.2) | 13.4 (1.2)
Statistical Analysis 1: Comparison: Add-on Citalopram Following Optimized Methylphenidate vs Add-on Placebo Following Optimized Methylphenidate; Test type: Superiority; p = 0.598, Multilevel growth curve model — priori threshold p<0.05; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-4.23 to 2.19]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected weekly during the study, including the 8th weeks of the trial.
Description: Adverse events were ascertained by checklists. These were completed by nurses (during inpatient admission) or parents (after discharge), all of whom were blind to treatment assignment, and instructed to rate what they observed without reference to changes from baseline irritability, time of day or severity of the presentation. Information on suicidality and manic symptoms were also routinely collected.
Arm/Group | Add-on Citalopram Following Optimized Methylphenidate | Add-on Placebo Following Optimized Methylphenidate
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 23/23 | 24/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Add-on Citalopram Following Optimized Methylphenidate (N=23) | Add-on Placebo Following Optimized Methylphenidate (N=26)
Dry mouth (Gastrointestinal disorders) | 3 | 4
Drooling (Gastrointestinal disorders) | 2 | 0
Increased thirst (Gastrointestinal disorders) | 3 | 3
Trouble swallowing (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 10 | 8
Vomiting (Gastrointestinal disorders) | 5 | 3
Stomach pains (Gastrointestinal disorders) | 13 | 16
Bloated abdomen (Gastrointestinal disorders) | 3 | 0
Changes in stool (Gastrointestinal disorders) | 8 | 6
Change in heart rate fast/slow (Cardiac disorders) | 1 | 2
Drowsiness morning/afternoon (Nervous system disorders) | 7 | 3
Dizziness (Nervous system disorders) | 5 | 1
Tiredness/fatigue (General disorders) | 12 | 9
Insomnia (General disorders) | 17 | 24
Early morning awakening (General disorders) | 3 | 3
Appetite changes (General disorders) | 23 | 21
Weight changes (General disorders) | 13 | 13
Fever (General disorders) | 1 | 3
Enuresis (Renal and urinary disorders) | 1 | 2
Eyes sensitive to light (Eye disorders) | 1 | 2
Headache (General disorders) | 11 | 12
Ringing or buzzing in ears (Ear and labyrinth disorders) | 0 | 2
Runny nose (General disorders) | 6 | 7
Easy bruising (General disorders) | 2 | 2
Anger (Psychiatric disorders) | 19 | 22
Agression (Psychiatric disorders) | 17 | 12
Nervousness (Psychiatric disorders) | 15 | 13
Clingy/separation anxiety (Psychiatric disorders) | 13 | 8
Loss of interest/apathy (Psychiatric disorders) | 7 | 6
Poor concentration (Psychiatric disorders) | 9 | 8
Disorganized thinking (Psychiatric disorders) | 2 | 1
Speech changes (Psychiatric disorders) | 7 | 6
Intrusiveness (Psychiatric disorders) | 17 | 15
Restless/Inability to sit still (Musculoskeletal and connective tissue disorders) | 16 | 19
Stiffness/Involuntary movements (Musculoskeletal and connective tissue disorders) | 2 | 5
Extreme stiffness/Lack of movement (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitches (Musculoskeletal and connective tissue disorders) | 1 | 2
Motor tics (Musculoskeletal and connective tissue disorders) | 8 | 11
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Severe or chronic cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Whezzing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash/itch (Skin and subcutaneous tissue disorders) | 8 | 5
Increased sweating (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Hair changes (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 4 | 1
Picking at skin or nails (Skin and subcutaneous tissue disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
The sample size was smaller than initially planned. Our primary measure of irritability Aberrant Behavior Checklist - Irritability subscale, did not prove suitable for the current study due to its design (i.e., different environments and informants)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT00794040/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT00794040/SAP_001.pdf